CLINICAL TRIAL: NCT04739462
Title: mHealth for Improvement of Access to Maternal Health Services in the Era of COVID-19 Pandemic (SMS Maama Project)
Brief Title: SMS Maama Project COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00010582
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Pregnancy Complications; Birth Injuries
MeSH Terms: conditions — Pregnancy Complications; Birth Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this arm will receive the study intervention.
  Interventions: Behavioral: mHealth Platform
- Routine Antenatal Care (No Intervention): Participants in this arm will receive no intervention.

INTERVENTIONS:
Behavioral: mHealth Platform — All participants randomized to the intervention group will receive 2-4 informational texts each week and will also receive interactive health screening questions throughout enrollment. A participant will also receive appointment reminder texts. All SMS text messages will be transmitted through a local organization known as The Medical Concierge Group (TMCG) via an electronic system that allows for bulk messaging. TMCG also staffs a 24-hour call line for those using TMCG services to call in for medical related questions. This call line is staffed by doctors and nurses; SMS Maama participants randomized to the interventional group will be able to access this call line free of charge as part of their enrollment in SMS Maama.
  Arms: Intervention

SUMMARY:
The study's purpose is to demonstrate the ability of an mHealth platform as a feasible way of sharing information in a time of restricted movement in order to inform future studies.

DETAILED DESCRIPTION:
The primary objective of this trial is to assess whether an mHealth platform increases maternal health knowledge in the areas of birth preparedness, pregnancy, and birth complications as measured by the pre- and post-surveys in comparison to routine antenatal care.

The secondary objectives of this trial are;

1. To provide knowledge of COVID-19 symptoms, transmission, diagnosis, and treatment, in a time of social distancing and learning.
2. To improve access and linkages to maternal health services and information as well as provide appropriate referrals for pregnant females.
3. Inform the adoption of mHealth into future health delivery plans.

ELIGIBILITY:
Inclusion Criteria:

* Own a personal mobile phone
* Attend ANC at Kisenyi Health Centre IV, Kawempe Hospital or Rubaga Hospital
* Are at least 24-26 weeks estimated gestational age
* Literate in English or Luganda
* Capable of sending/receiving text messages

Exclusion Criteria:

- Females who plan to travel out of Uganda during the study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Change in Pre- to Post-Intervention Knowledge | up to 18 weeks
  Outcome is reported as the percent of pregnant participants who recognize key danger signs during pregnancy, labor and childbirth, and postpartum period. Knowledge is measured pre-intervention (approximately 24-26 weeks gestation) and post-intervention (approximately 2 weeks following delivery). The timeframe is calculated to be 16-18 weeks.

SECONDARY OUTCOMES:
Change in Knowledge on COVID-19 | up to 18 weeks
  Outcome reported as the percent of pregnant participants who identify key symptoms, modes of transmission, and measures to prevent SARS-CoV-2 infection (COVID-19). Knowledge is measured pre-intervention (approximately 24-26 weeks gestation) and post-intervention (approximately 2 weeks following delivery). The timeframe is calculated to be 16-18 weeks.
Rate of COVID Testing | up to 18 weeks
  Outcome is reported as the percent of pregnant participants who were tested for SARS-CoV-2 during pregnancy.
Change in Pregnancy Risk Knowledge | up to 18 weeks
  Outcome is reported as the percent of pregnant participants who believe pregnant females are at increased risk for COVID-19. Knowledge is measured pre-intervention (approximately 24-26 weeks gestation) and post-intervention (approximately 2 weeks following delivery). The timeframe is calculated to be 16-18 weeks.
Change in Breastfeeding Knowledge | up to 18 weeks
  Outcome is reported as the percent of pregnant participants who believe it is safe to breastfeed their newborn if they have or have had COVID-19. Knowledge is measured pre-intervention (approximately 24-26 weeks gestation) and post-intervention (approximately 2 weeks following delivery). The timeframe is calculated to be 16-18 weeks.
Antenatal Care Rate | up to 18 weeks
  Outcome is reported as the percent of pregnant participants who attend at least 4 antenatal care visits.
Skilled Birth Attendance Rate | up to 18 weeks
  Outcome is reported as the percent of pregnant participants who give birth at a hospital.
Rate of Negative Pregnancy Outcomes | up to 18 weeks
  Outcome is reported as the percent of pregnant participants who experience a negative pregnancy outcome (e.g. maternal/neonatal complications, miscarriage, stillbirth, and/or neonatal death).

CONTACTS AND LOCATIONS:
Overall Officials: Betty Nakabuye, MBChB, MMed, Principal Investigator — Lubaga Hospital and School of Public Health, Makerere University; Jolly Beyeza, Principal Investigator — Mulago Specialised Women's Hospital and School of Medicine, Makerere University; Katelyn Pastick, Principal Investigator — University of Minnesota; Cheryl Robertson, Principal Investigator — University of Minnesota
Locations (2):
- University of Minnesota, Minneapolis, Minnesota, United States
- Makerere University, Kampala, Uganda